CLINICAL TRIAL: NCT06070545
Title: The Effect of Modified Supine Position on Urinary Elimination After Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esra Karagoz, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-66175679-514.99-1045359
Record Dates: First submitted 2023-09-06; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Urinary Retention
Keywords: Percutaneous Coronary Intervention; Patient Positioning; Urinary Elimination
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Modified supine position care
  Interventions: Other: Modified Supine Position
- Control Group (No Intervention): Standard Care

INTERVENTIONS:
Other: Modified Supine Position — Among the patients in the control group, for whom consent was obtained, the standard clinical procedure including supine after percutaneous coronary intervention (0 degrees flat on the back) will be provided, and for the patients in the experimental group, care including the modified supine position will be provided. The modified supine position is a position in which patients lie on their back with the head of the bed elevated at a 20-degree angle, with a pillow between the soles of their feet and the end of the bed. Both study groups will be required to lie supine in bed for 6 hours and stay in bed for 12 hours before ambulation is allowed in order not to increase the risk of local bleeding, as required by the clinical procedure.
  Arms: İntervention Group

SUMMARY:
Urinary retention is also a frequent complication after percutaneous coronary intervention applied via the femoral artery. The inability to manage this situation effectively leads to serious complications in the long term, prolonging the length of hospital stay and increasing the cost, as well as impairing the participants's comfort. In the investigators's country, no study has been found in which the effectiveness of an appropriate and effective lying position in performing urinary drainage in the bed in order to ensure urinary emptying and to minimize possible complications in participants undergoing percutaneous coronary intervention has been found. One study states that the modified supine position is an effective intervention on the amount of urine output in participants. In another study, it was determined that different degrees of bed height and position changes would be safe and effective in reducing regional pain and vascular complications (hematoma, bleeding, thrombosis, bruising, etc.). In this context, the aim of the study is to reveal the effect of the modified supine position on providing effective urinary drainage (hourly and 24-hour urine output) and preventing possible complications (urinary retention) in participants undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
Cardiovascular diseases are an important health problem in the world and in the investigators's country, and are among the leading causes of death in adults. According to the 2017 data of the Coronary Heart Disease and Risk Factors in Turkish Adults (TEKHARF) study, it is estimated that there are approximately 3.5 million coronary heart patients in the investigators country, this number increases by 4% per year in the investigators aging population, and 210 thousand individuals die from coronary heart disease annually.

Percutaneous coronary intervention is a revascularization method used in the treatment of coronary artery disease. Complications related to vascular access sites occur in 5-7% of patients undergoing percutaneous coronary intervention. The most common coronary vascular intervention complications are; hematoma, bleeding at the vascular access site, arterial pseudoaneurysm and arteriovenous fistula development. According to the latest guidelines and literature, bed rest ranges from 6 to 24 hours, especially after percutaneous coronary intervention applied via femoral route in order to prevent bleeding-related complications.

Another complication encountered after percutaneous coronary intervention applied through the femoral artery is difficulties in urinary drainage. Having long rest periods in the supine position and being able to urinate only in the supine position, without allowing knee bending, in order to prevent complications that may develop at the application site during this period; It can cause difficulty in emptying urine, incomplete emptying of the urine from the bladder, and retention.

In our country, no study has been found in which the effectiveness of an appropriate and effective lying position in performing urinary drainage in the bed in order to ensure urinary emptying and to minimize possible complications in patients undergoing percutaneous coronary intervention has been found. One study, states that the modified supine position is an effective intervention on the amount of urine output in patients. In another study, it was determined that different degrees of bed height and position changes would be safe and effective in reducing regional pain and vascular complications (hematoma, bleeding, thrombosis, bruising, etc.). In this context, the aim of the study is to reveal the effect of the modified supine position on providing effective urinary drainage (hourly and 24-hour urine output) and preventing possible complications (urinary retention) in patients undergoing percutaneous coronary intervention.

Formation of the Experimental Group and Interventions:

Written and verbal consent will be obtained from participants who agree to participate in the study. Among the participants in the control group, for whom consent was obtained, the standard clinical procedure including supine after percutaneous coronary intervention (0 degrees flat on the back) will be provided, and for the participants in the experimental group, care including the modified supine position will be provided. The modified supine position is a position in which participants lie on their back with the head of the bed elevated at an angle of 20 degrees, with a pillow between the soles of their feet and the end of the bed. Both study groups will be required to lie supine in bed for 6 hours and stay in bed for 12 hours before ambulation is allowed in order not to increase the risk of local bleeding, as required by the clinical procedure. For this reason, these measurements determined for urinary excretion will be followed by the investigator for 6 hours. In addition, participants in the experimental and control groups will be encouraged to drink and urinate within 2 hours after percutaneous coronary intervention in order to facilitate the elimination of contrast material, and the amount of fluid ingested and excreted for 6 hours will be recorded by the investigator. The primary outcome variables of the study in determining bladder function will be time to first urgency and voiding function. participants with the feeling of urination will call the investigative nurse with the call bell and the time will be followed from the moment the slider/duck/voiding bottle is placed until the end of urination. This time will give the first urination time and will be evaluated at 4 levels. These 4 levels; Level 0: Urinating within 1 minute Level 1: Urinating within 1 to 30 minutes Level 2: Urinating within 1 to 30 minutes and needing assistance such as massage or heat pack to do so Level 3: Self or other It is stated that he cannot urinate with help methods and needs a urinary catheter. Levels 2 to 3 are considered impaired voiding. Secondary research variables are initial voiding volume and assessment of urinary retention volume. The first voiding volume will be measured, and for urinary retention, the volume of urine remaining in the bladder will be measured and recorded with a portable ultrasound device. For this measurement, the investigator nurse nurse will receive training on how to measure the volume of urine remaining in the bladder with an ultrasound device. The need for catheterization within the first 24 hours after percutaneous coronary intervention will be defined as urinary retention.

To evaluate the safety of the modified supine position, the presence/absence of complications such as back pain, deep vein thrombosis, hematoma, ecchymosis and pseudoaneurysm that may develop after percutaneous coronary intervention will be recorded. Pain; Before and immediately after the procedure, participants will be assessed by the Visual Analogue Scale (VAS) for pain at the puncture site or back. Anxiety will be measured as they are risk factors for post-intervention urinary retention. In addition, anxiety levels will be evaluated before the procedure in order to ensure conjugation in the experimental and control groups. Vascular intervention complications such as thrombosis, hematoma, ecchymosis and pseudoaneurysm will be observed for 6 hours and recorded in case of change. The dorsalis pedis pulse, foot color and temperature change will be evaluated to detect thrombosis. In addition, the bladder diary (voiding/day, nocturia/day, time between voiding-min, mean voiding volume-ml) and the amount of fluid ingested and excreted during the discharge of the participants will be given by the investigator 24 hours after the procedure by phone monitoring. The participant will provide training to the participant and his or her relatives who are primarily responsible for their care in filling out this diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cardiovascular disease,
* Elective hospitalizations and transfemoral percutaneous coronary intervention,
* Ability to urinate without problems and express the desire to urinate,
* Able to communicate verbally,
* Not having any disability in terms of consciousness and sensory organs (Mini Mental Score 25 and above),
* Adult patients who volunteer to participate in the study will be included.

Exclusion Criteria:

•Participants who underwent intraoperative foley catheterization, who had a history of prostate hyperplasia, prostate carcinoma, urinary tract infection, urological disease, sensory disorders or neurological problems, who had the procedure performed under spinal or epidural anesthesia, who cannot tolerate the supine position according to the clinical procedure, and who cannot communicate in Turkish will not be included.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time taken to reach first voiding function. | Measurement of the time from the moment the bedpan/duck/urine bottle was placed to the end of urination in participants who felt the urge to urinate within the first 6 hours after coronary angiography.
  This time will give the first urination time and will be evaluated at 4 levels. These 4 levels; Level 0: Urinating within 1 minute, Level 1: Urinating within 1 to 30 minutes, Level 2: Urinating within 1 to 30 minutes and needing assistance such as massage or heat pack to do so, Level 3: Unable to urinate by self or other means of assistance and needs a urinary catheter. Levels 2 to 3 are considered impaired voiding.
Standardized Mini Mental State Examination (SMMSE) | İmmediately before percutaneous coronary intervention, baseline.
  SMMSE scores of 23 and below are considered to be indicative of cognitive impairment. In this study, patients with 25 points and above will be included in the study.

SECONDARY OUTCOMES:
It is the evaluation of initial voiding volume and urinary retention volume. | Immediately after first urination.
  The first voiding volume will be measured, and for urinary retention, the volume of urine remaining in the bladder will be measured and recorded with a portable ultrasound device.
Change in pain as measured by Visual Analog Scale. | İmmediately before percutaneous coronary intervention and immediately after the first voiding.
  Measured using the Visual Analog Scale for pain, on a scale of 0 to 10, in which a higher score means an increased level of pain.
Change in anxiety as measured by Visual Analog Scale (VAS-A). | İmmediately before percutaneous coronary intervention and immediately after the first voiding.
  Measured using the Visual Analog Scale for anxiety, on a scale of 0 to 10, in which a higher score means an increased level of anxiety.
Evaluation of the presence of thrombosis in the extremity where the femoral artery is located where percutaneous coronary intervention is performed. | The first 6 hours after the procedure.
  The presence of thrombosis will be accepted if at least one of the following conditions is present: absence of dorsalis pedis pulse, cyanosis of the extremity, increase in extremity diameter and temperature.
Follow-up of post-procedure fluid intake and urine output as measured by the European Association of Urology bladder diary. | From the 6th hour to the 24th hour after the procedure.
  The European Association of Urology bladder diary includes information about the participant's hourly fluid intake, urine output, and urination characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdollahi AA, Mehranfard S, Behnampour N, Kordnejad AM. Effect of Positioning and Early Ambulation on Coronary Angiography Complications: a Randomized Clinical Trial. J Caring Sci. 2015 Jun 1;4(2):125-34. doi: 10.15171/jcs.2015.013. eCollection 2015 Jun. PMID 26171374
- [Background] Açıkel S, Atar İ, Bozbaş H, Aydınalp A, Bilgi M, Yıldırır A, Özin B ve Müderrisoğlu H. TGKD Femoral bölgede hematom. 2010; 14(3):11-116.
- [Background] Alagöl B. İdrar retansiyonu: Üroloji 3. Baskı; Ed.: Osman İnci. Ankara: Güneş Kitabevi 2006; 1-5.
- [Background] Bakan G. Perkütan koroner girişimlerde kanıta dayalı bakım uygulamaları. Turkish Journal of Cardiovascular Nursing. June 2016; 7(sup 1):26-34.
- [Background] Liu YS, Wei S, Elliott M. The effects of a catheter clamping protocol on bladder function in neurosurgical patients: a controlled trial. Int J Nurs Pract. 2015 Feb;21(1):29-36. doi: 10.1111/ijn.12209. Epub 2013 Nov 13. PMID 24219753
- [Background] Liu Y, Zhang Y, Wu Y, Elliott M. A Modified Supine Position Facilitates Bladder Function in Patients Undergoing Percutaneous Coronary Intervention: A Randomized Controlled Clinical Trial. J Cardiovasc Nurs. 2018 Mar/Apr;33(2):152-159. doi: 10.1097/JCN.0000000000000436. PMID 28723835
- [Background] Mohammady M, Atoof F, Sari AA, Zolfaghari M. Bed rest duration after sheath removal following percutaneous coronary interventions: a systematic review and meta-analysis. J Clin Nurs. 2014 Jun;23(11-12):1476-85. doi: 10.1111/jocn.12313. Epub 2013 Sep 13. PMID 24028631
- [Background] Onat A. TEKHARF 2017 Tıp dünyasının kronik hastalılarına öncülük. Erişim Adresi: https://file.tkd.org.tr/PDFs/TEKHARF-2017.pdf. Erişim Tarihi: 25.06.2022.
- [Background] Niknam Sarabi H, Farsi Z, Butler S, Pishgooie AH. Comparison of the effectiveness of position change for patients with pain and vascular complications after transfemoral coronary angiography: a randomized clinical trial. BMC Cardiovasc Disord. 2021 Feb 25;21(1):114. doi: 10.1186/s12872-021-01922-w. PMID 33632127
- [Background] Türk kardiyoloji derneği girişimsel kardiyolojide yetkinlik kılavuzu. Erişim Adresi: https://tkd.org.tr/kilavuz/girisimsel_kilavuz.htm. Erişim Tarihi: 26.06.2022.
- [Background] Uslu Y ve Yavuz M. Ameliyat sonrası üriner retansiyon ve yönetimi. Yeni Üroloji Dergisi - The New Journal of Urology. 2016; 11(1):48-53.